CLINICAL TRIAL: NCT04679909
Title: A Phase 1, Double-blind, Randomized, Placebo-controlled, First-in-Human Study of the Safety and Immunogenicity of AdCOVID Administered as One or Two Doses
Brief Title: Safety and Immunogenicity of AdCOVID in Healthy Adults (COVID-19 Vaccine Study)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Altimmune, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ALT-501-101
Record Dates: First submitted 2020-12-21; First posted 2020-12-22 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Healthy Volunteers
Keywords: COVID-19; SARS-CoV-2; Intranasal Vaccine
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Single Low Dose AdCOVID (Experimental)
  Interventions: Biological: AdCOVID
- Single Medium Dose AdCOVID (Experimental)
  Interventions: Biological: AdCOVID
- Single High Dose AdCOVID (Experimental)
  Interventions: Biological: AdCOVID
- Two Low Doses AdCOVID (Experimental)
  Interventions: Biological: AdCOVID
- Two Medium Doses AdCOVID (Experimental)
  Interventions: Biological: AdCOVID
- Two High Doses AdCOVID (Experimental)
  Interventions: Biological: AdCOVID
- Single Dose Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- Two Dose Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: AdCOVID — Administered intranasally
  Arms: Single High Dose AdCOVID; Single Low Dose AdCOVID; Single Medium Dose AdCOVID; Two High Doses AdCOVID; Two Low Doses AdCOVID; Two Medium Doses AdCOVID
Other: Placebo — Administered intranasally
  Arms: Single Dose Placebo; Two Dose Placebo

SUMMARY:
A study to evaluate the immune response and safety of AdCOVID administered as an intranasal spray in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ages 18 to 55 years, inclusive
* Good general health status
* Screening laboratory results within institutional normal range or Grade 1 abnormality if the Investigator documents clinical insignificance. Grade 2 laboratories may be permissible if considered not clinically significant by the investigator.
* For women who have not been surgically sterilized or who do not have laboratory confirmation of postmenopausal status, negative pregnancy test
* Willingness to practice a highly effective method of contraception
* Ability and willingness to comply with all aspects of the study, including nasopharyngeal swabs and blood and urine samples, through the entire study period

Exclusion Criteria:

* Subjects at increased risk of exposure to SARS-CoV-2, including healthcare workers, emergency response personnel, and those with known contact with COVID-19 patients
* Pregnant or lactating women or planning to conceive a child during the next 3 months
* Body mass index (BMI) > 30.0 kg/m2
* Acute COVID-19, a positive test result for SARS-CoV2 infection, a positive SARS-CoV-2 serology for prior SARS-CoV-2 infection at screening, or exposure within 14 days to an individual with acute COVID-19
* An acute respiratory illness
* Positive result for HIV, hepatitis B virus, or hepatitis C virus at screening
* Chronic or current cigarette smoking
* Any medical, psychiatric, or social condition or occupational or other responsibility that in the judgment of the Investigator would interfere with or serve as a contraindication to protocol adherence, assessment of safety (including reactogenicity), or a subject's ability to give informed consent

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-12-21 (Actual)

PRIMARY OUTCOMES:
Reactogenicity | For 7 days after vaccination
  Counts and percentages of subjects with local and systemic events
Adverse Events (AEs) | Day 1 to Day 57
  Counts and percentages of subjects with AEs

SECONDARY OUTCOMES:
Anti-SARS-CoV-2 spike IgG antibody levels | Day 1 to Day 366
Neutralizing antibody titer against live and/or pseudotyped SARS-CoV-2 virus | Day 1 to Day 366

OTHER OUTCOMES:
Anti-SARS-CoV-2 RBD T cell responses by interferon (IFN)-gamma enzyme-linked immunosorbent spot (ELISpot) | Day 1 to Day 366
Mucosal antibody responses in nasopharyngeal swabs (anti-SARS-CoV-2 spike IgA titers) | Day 1 to Day 366

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - AGA Clinical Trials, Hialeah, Florida
  - Optimal Research, Melbourne, Florida
  - Optimal Research, Peoria, Illinois
  - Optimal Research, Rockville, Maryland
  - Optimal Research, Austin, Texas
  - Clinical Trials of Texas, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No